CLINICAL TRIAL: NCT00116402
Title: A Pilot Study of the Mechanism of Synergism Between Fluticasone (FP) and Salmeterol in Preventing Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Brief Title: A Pilot Study of the Mechanism of Synergism Between FP and Salmeterol in Preventing COPD Exacerbations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13426B
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Chronic Obstructive; Pulmonary Disease; Inhaled Corticosteroids; Airway Inflammation; Bronchoscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): will start with fluticasone 220 mcg BID first and then crossover to combination therapy with salmeterol 50 mcg BID
  Interventions: Drug: fluticasone and salmeterol
- 2 (Active Comparator): salmeterol 50 mcg BID then crossover to combination therapy with fluticasone 220 mcg BID
  Interventions: Drug: fluticasone and salmeterol

INTERVENTIONS:
Drug: fluticasone and salmeterol — 1. will start with fluticasone 220 mcg BID first and then crossover to combination therapy with salmeterol 50 mcg BID
  2. will start with salmeterol 50 mcg BID first and then crossover to combination therapy with fluticasone 220 mcg BID.

SUMMARY:
The purpose of this study is to evaluate the blood and airway of subjects with mild to moderate COPD while undergoing standard treatment.

DETAILED DESCRIPTION:
Our objective is to examine the mechanism of the additive/synergistic properties of b2-adrenoceptor stimulation and corticosteroid receptor activation in:

* Preventing neutrophil adhesion to specific endothelial ligands, e.g. ICAM-1 and
* Undergoing activation as a consequence of this adhesion.

We hypothesize that combination therapy with salmeterol + fluticasone (FP) will:

* Augment the inhibition of adhesion of neutrophils obtained from the peripheral blood of study subjects in vitro, by blocking gIV-PLA2 translocation to the nuclear membrane as for eosinophils;
* Augment the inhibition of transendothelial migration of neutrophils into airways of subjects with chronic obstructive pulmonary disease;
* Augment the numbers and concentrations of pro-inflammatory products in the bronchoalveolar lavage fluid; and
* Decrease the number of neutrophils in the bronchial tissue of endobronchial biopsies of treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 50 years of age
* Physiologic evidence of COPD defined per ATS guidelines as: cigarette smoking history >20 pack years, FEV1/FVC <70%
* Patients must have a post-bronchodilator FEV1 >50% of predicted value at enrollment
* Patient must have an O2 saturation measure by pulse oximetry >90% on RA
* Must be able to participate in the study, willing to give informed consent, and comply with the study restrictions

Exclusion Criteria:

* Women of child-bearing potential defined as females who are less than 5 years post menopausal unless they have had a hysterectomy or bilateral oophorectomy
* Observation of any solitary nodule in the lung requiring further medical intervention
* Patients on maintenance therapy with oral steroids
* Patients with giant bullous disease
* Significant other medical conditions, which in the opinion of the investigator, will interfere with the patient's ability to perform the study tests
* Presence of a coagulopathy as defined by a platelet count <100,000/mm3, and PT and PTT >1.2 x the upper limit of normal
* Concurrent enrollment or participation in any other clinical trials within the past 30 days
* Primary diagnosis of asthma
* History of alpha 1 antitrypsin deficiency
* Any clinically significant and active pulmonary disease that could contribute to dyspnea
* Current systemic and inhaled steroids and theophylline

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-01; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To evaluate blood and airway neutrophil population in COPD patients by examining adhesion and migration in patients with mild to moderate COPD | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Imre Noth, M.D., Principal Investigator — University of Chicago
Locations (1):
- Department of Medicine, Pulmonary & Critical Care Section, The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Soriano JB, Kiri VA, Pride NB, Vestbo J. Inhaled corticosteroids with/without long-acting beta-agonists reduce the risk of rehospitalization and death in COPD patients. Am J Respir Med. 2003;2(1):67-74. doi: 10.1007/BF03256640. PMID 14720023
- [Background] Hanania NA, Darken P, Horstman D, Reisner C, Lee B, Davis S, Shah T. The efficacy and safety of fluticasone propionate (250 microg)/salmeterol (50 microg) combined in the Diskus inhaler for the treatment of COPD. Chest. 2003 Sep;124(3):834-43. doi: 10.1378/chest.124.3.834. PMID 12970006
- [Background] Hattotuwa KL, Gizycki MJ, Ansari TW, Jeffery PK, Barnes NC. The effects of inhaled fluticasone on airway inflammation in chronic obstructive pulmonary disease: a double-blind, placebo-controlled biopsy study. Am J Respir Crit Care Med. 2002 Jun 15;165(12):1592-6. doi: 10.1164/rccm.2105025. PMID 12070058
- [Background] Kim KP, Rafter JD, Bittova L, Han SK, Snitko Y, Munoz NM, Leff AR, Cho W. Mechanism of human group V phospholipase A2 (PLA2)-induced leukotriene biosynthesis in human neutrophils. A potential role of heparan sulfate binding in PLA2 internalization and degradation. J Biol Chem. 2001 Apr 6;276(14):11126-34. doi: 10.1074/jbc.M004604200. Epub 2000 Dec 15. PMID 11118430
- [Background] Kim YJ, Kim KP, Han SK, Munoz NM, Zhu X, Sano H, Leff AR, Cho W. Group V phospholipase A2 induces leukotriene biosynthesis in human neutrophils through the activation of group IVA phospholipase A2. J Biol Chem. 2002 Sep 27;277(39):36479-88. doi: 10.1074/jbc.M205399200. Epub 2002 Jul 17. PMID 12124392
- [Background] Chang PS, Absood A, Linderman JJ, Omann GM. Magnetic bead isolation of neutrophil plasma membranes and quantification of membrane-associated guanine nucleotide binding proteins. Anal Biochem. 2004 Feb 15;325(2):175-84. doi: 10.1016/j.ab.2003.10.039. PMID 14751252
- [Background] Myou S, Zhu X, Boetticher E, Myo S, Meliton A, Lambertino A, Munoz NM, Leff AR. Blockade of focal clustering and active conformation in beta 2-integrin-mediated adhesion of eosinophils to intercellular adhesion molecule-1 caused by transduction of HIV TAT-dominant negative Ras. J Immunol. 2002 Sep 1;169(5):2670-6. doi: 10.4049/jimmunol.169.5.2670. PMID 12193740
- [Background] Reumaux D, de Boer M, Meijer AB, Duthilleul P, Roos D. Expression of myeloperoxidase (MPO) by neutrophils is necessary for their activation by anti-neutrophil cytoplasm autoantibodies (ANCA) against MPO. J Leukoc Biol. 2003 Jun;73(6):841-9. doi: 10.1189/jlb.1102567. PMID 12773517
- [Background] Zhu X, Munoz NM, Kim KP, Sano H, Cho W, Leff AR. Cytosolic phospholipase A2 activation is essential for beta 1 and beta 2 integrin-dependent adhesion of human eosinophils. J Immunol. 1999 Sep 15;163(6):3423-9. PMID 10477614
- [Background] Meliton AY, Munoz NM, Liu J, Lambertino AT, Boetticher E, Myo S, Myou S, Zhu X, Johnson M, Leff AR. Blockade of LTC4 synthesis caused by additive inhibition of gIV-PLA2 phosphorylation: Effect of salmeterol and PDE4 inhibition in human eosinophils. J Allergy Clin Immunol. 2003 Aug;112(2):404-10. doi: 10.1067/mai.2003.1637. PMID 12897749
- [Background] Reid DW, Ward C, Wang N, Zheng L, Bish R, Orsida B, Walters EH. Possible anti-inflammatory effect of salmeterol against interleukin-8 and neutrophil activation in asthma in vivo. Eur Respir J. 2003 Jun;21(6):994-9. doi: 10.1183/09031936.03.00109702. PMID 12797494
- [Background] Qiu Y, Zhu J, Bandi V, Atmar RL, Hattotuwa K, Guntupalli KK, Jeffery PK. Biopsy neutrophilia, neutrophil chemokine and receptor gene expression in severe exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2003 Oct 15;168(8):968-75. doi: 10.1164/rccm.200208-794OC. Epub 2003 Jul 11. PMID 12857718